CLINICAL TRIAL: NCT03136081
Title: IMMUNOCANDIDA Candida Host Defense Response After Septic Shock in the Critically Ill
Brief Title: Candida Host Defense Response After Septic Shock in the Critically Ill
Acronym: IMMUNOCANDIDA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF 9358
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Septic Shock; Candidiasis
Keywords: Septic shock; Candidiasis; Candidemia; Bacteremia; Immunoparalysis
MeSH Terms: conditions — Shock, Septic; Candidiasis; Candidemia; Bacteremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — It will be simply about additional tubes taken during the taking of the day blood, usually realized on the catheter thus without pain nor risk of bruise. We also préleverons one sample of urine every 2 days for analysis of laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Septic shock and candidiasis: The realized analyses will be two types:
  1/an immunological analysis that is the characterization of the capacities of defense against germs and 2/a search(research) of Candida by microscopic examination and culture on circles of growth but also the research for the genome of the mushroom by a state-of-the-art technique of the laboratory of mycology ( PCR). Usual takings of research for bacteria.
  Interventions: Diagnostic Test: Candidiasis infection occurence

INTERVENTIONS:
Diagnostic Test: Candidiasis infection occurence — Candidiasis infection occurence

SUMMARY:
Septic shock is associated with acquired immunoparalysis which is associated with a high risk of nosocomial acquired infection. Nosocomial candidiasis is associated with a 50% rate of mortality but is difficult to diagnose. The use of colonization indexes and risk factors on the other hand expose to unnecessary use of antifungals. The aim of the present study is to evaluate whether the host response to infection associated with candida biomarkers would help to anticipate the candidiasis onset.

DETAILED DESCRIPTION:
Single center prospective observationnal study. Inclusion: all consecutive patients subsequently to a septic shock with no Candida infection.

Measured parameters: host response (HLADR, CD64, inflammatory cytokines consecutive to LPS exposition) and Candida biomarkers (beta D Glucan, Mannan Ag and Ig), demographics, outcome (occurence of Candida nosocomial infection, morbidity and survival)

ELIGIBILITY:
Inclusion Criteria:

Age > = 18 years

* The patients in toxic shock defined according to the Bone criteria
* Informed consent of the patient or his reliable person (poursuit consent in this case). Possibility of inclusion according to the emergency procedure with the obligation of research for the consent with the reliable person and with the patient.
* Obligation of membership or beneficiary to have a national insurance

Exclusion Criteria:

* Pregnant or breast-feeding women according to the article L1121-5 of the CSP
* Vulnerable people according to the article L1121-6 of the CSP 9358 _ "
* Neutropénie 500 / mm3
* Infection by the HIV, the hepatitis C or B active column
* Biotherapics (anti-CD20, anti-TNFa, anti-IL-6)
* Treatments immunosuppresseurs (methotrexate, azathioprine, cyclophosphamide, mycophenolate mofétil, cyclosporine, tacrolimus)
* Corticosteroid therapy = 1mg / kg of equivalent prednisone for more than a month
* Toxic shock due to a deep candidiasis in the admission in resuscitation
* Congenital deficits of Th17 (cutanéo-mucous candidiasis chronicles, syndrome of hyper IgE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all consecutive patients subsequently to a septic shock with no Candida infection.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Candidiasis infection occurence | Day 28 survival
  Outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital St Eloi, Montpellier, France

IPD SHARING:
Plan to Share IPD: No